CLINICAL TRIAL: NCT06043804
Title: Study on Doppler Ultrasound Measurement of Changes in Uterine Artery Blood Flow in Normal First Trimester Pregnancies and Its Prediction on Abortion
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2023-07-208
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Abnormal Uteroplacental Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pregnant woman: healthy pregnant woman
  Interventions: Other: Doppler ultrasound measurement of changes in uterine artery blood flow
- Pregnant women with recurrent pregnancy loss: Spontaneous abortion of three or more consecutive sexual partners
  Interventions: Other: Doppler ultrasound measurement of changes in uterine artery blood flow

INTERVENTIONS:
Other: Doppler ultrasound measurement of changes in uterine artery blood flow — Doppler ultrasound measurement of changes in uterine artery blood flow

SUMMARY:
Objective:To explore the study of Doppler ultrasound in first trimester pregnancies to measure the change of uterine artery blood flow in normal pregnancies and the prediction on abortion, which provides a certain reference for the change trend of uterine artery blood flow in normal first trimester pregnancies and the prediction of Doppler ultrasound measurement in abortion.

Method:Pregnant women who underwent natural conception and single birth prenatal examination in the Obstetrics Department of the Second Affiliated Hospital of Wenzhou Medical University from October 1, 2023 to December 31, 2025 were selected as the study population. Eligible women were preliminarily screened according to the inclusion conditions of the study objects, and basic information of women in each group was compared: Maternal age, gestational time, birth time, gestational week, abortion history, maternal BMI, maternal MAP, smoking status, serum HCG, subchorionic hematoma, fetal bradycardia, left and right uterine aorta pulse index (PI), resistance index (RI) and systolic/diastolic ratio (S/D), etc. To investigate the effect of Doppler ultrasonography on the measurement of uterine artery blood flow in normal pregnancy and the prediction of abortion.

ELIGIBILITY:
Healthy pregnant women Group

Inclusion Criteria:

1. Intrauterine pregnancy sac and cardiac activity were confirmed by ultrasound examination at 6 weeks;
2. Complete maternal clinical data;

Exclusion Criteria:

1. The level of chorionic gonadotropin (HCG) was static or decreased by ultrasonography;
2. multiple pregnancy;
3. Patients with congenital uterine malformations, uterine fibroids and any other uterine disease;
4. Patients who have chronic diseases or are receiving chronic treatment.

Pregnant women with recurrent pregnancy loss Group

Inclusion Criteria:

1. Intrauterine pregnancy sac and cardiac activity were confirmed by ultrasound examination at 6 weeks;
2. Complete maternal clinical data;
3. There has been a history of spontaneous abortion with the same sexual partner for two or more consecutive times;

Exclusion Criteria:

1. The level of chorionic gonadotropin (HCG) was static or decreased by ultrasonography;
2. multiple pregnancy;
3. Patients with congenital uterine malformations, uterine fibroids and any other uterine disease;
4. Patients who have chronic diseases or are receiving chronic treatment.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pulsatility index | it can be monitored for up to 12 weeks
  Pulsatility index of the left and right main uterine arteries
Resistive index | it can be monitored for up to 12 weeks
  Resistive index of the left and right main uterine arteries
Systolic-to-diastolic ratio | it can be monitored for up to 12 weeks
  Systolic-to-diastolic ratio of the left and right main uterine arteries